CLINICAL TRIAL: NCT02682680
Title: Goal Achievement of A1c and LDL in a Randomized Trial Comparing Colesevelam vs. Ezetimibe as Add-on to Baseline Statin Therapy: The GOAL-RCT Trial
Brief Title: Randomized Trial Comparing Colesevelam vs. Ezetimibe
Acronym: GOAL-RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Harpreet Bajaj, Endocrinologist, LMC Diabetes & Endocrinology Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOAL RCT
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; hyperlipidaemia; colesevelam; ezetimibe; LDL cholesterol; glycated hemoglobin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperlipidemias | interventions — Colesevelam Hydrochloride; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colesevelam (Experimental): Colesevelam 3.75 g daily (tablets or oral suspension) for 24 weeks
  Interventions: Drug: Colesevelam
- Ezetimibe (Active Comparator): Ezetimibe 10 mg once daily for 24 weeks
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Colesevelam — Colesevelam 3.75 g daily for 24 weeks
  Other Names: Lodalis; Welchol
  Arms: Colesevelam
Drug: Ezetimibe — Ezetimibe 10 mg daily for 24 weeks
  Other Names: Ezetrol; Zetia
  Arms: Ezetimibe

SUMMARY:
A 24-week, randomized, open-label study investigating the efficacy, safety and tolerability of colesevelam 3.75 g daily compared to ezetimibe 10 mg daily, as an add-on to baseline statin therapy in patients with type 2 diabetes mellitus (T2DM) who are not at target for glycated hemoglobin (HbA1c) (> 7.0%) and low-density lipoprotein (LDL) cholesterol (> 2.0 mmol/L).

DETAILED DESCRIPTION:
This study will enroll 200 adult patients with T2DM who are not at target for HbA1c and LDL cholesterol. Patients who are on baseline statin therapy will be randomly assigned in a 1:1 ratio to colesevelam 3.75 g daily for 24 weeks, or ezetimibe 10 mg daily for 24 weeks. If a patient has statin intolerance, they may be on a fibrate and/or niacin, or on no lipid lowering therapy. The primary efficacy objectives are

1. to demonstrate that colesevelam 3.75 g daily is non-inferior to ezetimibe 10 mg daily as add-on to statin therapy for patients achieving a composite target of HbA1c (≤ 7.0%) and LDL cholesterol (≤ 2.0 mmol/L) at week 24, and
2. to compare the proportion of patients achieving a composite target of HbA1c (≤ 7.0%) and LDL cholesterol (≤ 2.0 mmol/L) at week 24.

This study will also assess the primary composite outcome in a sub-group of patients on sodium/glucose cotransporter 2 inhibitor (SGLT2i) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes > 6 months
2. HbA1c level between 7.1 to 10.0% (inclusive) within three months of study enrollment
3. LDL cholesterol > 2.0 mmol/L within three months of study enrollment
4. Receiving a stable dose of statin for a minimum of three months, which the investigator does not plan to change over the 24-week trial period. If patient has documented statin intolerance, may be on a fibrate and/or niacin, or on no lipid lowering therapy
5. Stable diabetes medications for previous three months (apart from adjustment of insulin dose)
6. Informed consent

Exclusion Criteria:

1. Use of a second lipid lowering therapy other than statin within three months of study enrolment, unless on a fibrate and/or niacin if patient has statin intolerance
2. Triglycerides ≥ 5.0 mmol/L or incalculable LDL cholesterol
3. Significant liver enzyme or CK elevation defined as CK or ALT ≥ 3x upper limit of normal (ULN)

5) Pregnant or breast feeding or planning to become pregnant or breast feed during the study 6) Chronic kidney disease (CKD) stage ≥4 or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m-squared 7) Severe gastroparesis or history of significant bowel resection 8) Current use of any Investigational Product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve target HbA1c and LDL cholesterol | 24 weeks
  target HbA1c: ≤ 7.0%; target LDL cholesterol: ≤ 2.0 mmol/L

SECONDARY OUTCOMES:
Proportion of subjects who achieve the primary outcome measure in the sub-group of subjects on sodium/glucose cotransporter 2 inhibitor (SGLT2i) therapy | 24 weeks
Absolute change in LDL cholesterol | 24 weeks
Absolute change in non-high-density lipoprotein (non-HDL) cholesterol | 24 weeks
Absolute change in fasting plasma glucose (FPG) | 24 weeks
Absolute change in HbA1c | 24 weeks
Absolute change in LDL cholesterol in sub-group of subjects on SGLT2i therapy | 24 weeks
Absolute change in non-HDL cholesterol in sub-group of subjects on SGLT2i therapy | 24 weeks
Absolute change in FPG in sub-group of subjects on SGLT2i therapy | 12 weeks and 24 weeks
Absolute change in HbA1c in sub-group of subjects on SGLT2i therapy | 12 weeks and 24 weeks
Proportion of subjects achieving a composite target of glycemic control, LDL cholesterol control and blood pressure control | 24 weeks
  glycemic control: A1c ≤ 7.0%; LDL cholesterol control: ≤ 2.0 mmol/L; blood pressure control: ≤ 130/80 mm Hg
Proportion of subjects achieving a composite target of glycemic control with no hypoglycemia and no weight gain | 24 weeks
Proportion of subjects with ≥ 0.3% reduction in HbA1c and ≥ 10% reduction in LDL cholesterol from baseline | 24 weeks
Proportion of subjects with ≥ 0.5% reduction in HbA1c and ≥ 15% reduction in LDL cholesterol | 24 weeks
Absolute change in high-sensitivity C-reactive protein (hs-CRP) levels from baseline | 24 weeks
Absolute change in triglyceride levels from baseline | 24 weeks
Proportion of subjects achieving target HbA1c and LDL cholesterol in the sub-group of subjects on non-insulin therapies | 24 weeks
Absolute change in FPG in the sub-group of subjects on non-insulin therapies | 24 weeks
Absolute change in HbA1c in the sub-group of subjects on non-insulin therapies | 24 weeks
Absolute change in LDL cholesterol in the sub-group of subjects on non-insulin therapies | 24 weeks
Absolute change in non-HDL cholesterol in the sub-group of subjects on non-insulin therapies | 24 weeks
Rate of non-severe and severe hypoglycemia | 24 weeks
  Severe hypoglycemia is defined as hypoglycemia requiring third party intervention of another person to actively administer carbohydrate, glucagon or other resuscitative actions.
Absolute change in alanine aminotransferase (ALT) | 24 weeks
Absolute change in creatine kinase (CK) | 24 weeks

OTHER OUTCOMES:
Change in body weight | 24 weeks
Change in body mass index (BMI) | 24 weeks
Change in waist circumference | 24 weeks
Effect of colesevelam versus ezetimibe on the increased LDL cholesterol levels typically observed with initiation of SGLT2i therapy | 24 weeks
Persistence of therapy of colesevelam versus ezetimibe | 24 weeks
Persistence of therapy of colesevelam versus ezetimibe in the sub-group of subjects on SGLT2i therapy | 24 weeks
Mean dose of colesevelam | 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harpreet Bajaj, MD, Principal Investigator — LMC Diabetes & Endocrinology
Locations (9):
- Canada (9):
  - LMC Calgary, Calgary, Alberta
  - LMC Barrie, Barrie, Ontario
  - LMC Brampton, Brampton, Ontario
  - LMC Etobicoke, Etobicoke, Ontario
  - LMC Markham, Markham, Ontario
  - LMC Oakville, Oakville, Ontario
  - LMC Thornhill, Thornhill, Ontario
  - Manna Toronto, Toronto, Ontario
  - LMC Bayview, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No